CLINICAL TRIAL: NCT05450315
Title: Effects of Targeted Versus Generic Print Materials on Physical Activity and Quality of Life in Young Adult Cancer Survivors: A Randomized Control Trial
Brief Title: Targeted Vs Generic Print Materials on Physical Activity and Quality of Life in Young Adult Cancer Survivors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S2Survive
Record Dates: First submitted 2015-05-26; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2018-10

CONDITIONS: Behaviour Change
Keywords: Physical Activity; Young Adult Cancer; Behavior Change
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TARG (Experimental): Group will receive physical activity information targeted to young adult cancer survivors
  Interventions: Behavioral: Stride to Survive:An Exercise Guide for Young Adult Cancer Survivors
- CPAG (Active Comparator): Group will receive the Canadian Public Health Guidelines
  Interventions: Behavioral: Canadian Physical Activity Guidelines

INTERVENTIONS:
Behavioral: Stride to Survive:An Exercise Guide for Young Adult Cancer Survivors
  Arms: TARG
Behavioral: Canadian Physical Activity Guidelines
  Arms: CPAG

SUMMARY:
Young adult cancer survivors (YACS) are an understudied group in cancer survivorship research that have unique psychosocial, medical and survivorship issues. Physical activity (PA) has important effects on health-related outcomes in middle-aged and older cancer survivors and preliminary research suggests similar benefits in YACS (18-39 years). Unfortunately, only about half of YACS report meeting public health PA guidelines and there are no interventions or resources available to help YACS increase their PA. The purpose of this study is to test a physical activity guidebook that was developed for YACS based on the theory of planned behavior (TPB). The PA guidebook will be evaluated in a randomized controlled trial. Specifically, 300 YACS will be randomly assigned to (a) Canada's PA guidelines for adults or (b) the YACS PA guidebook. YACS will complete assessments of PA, quality of life, and psychosocial variables at baseline (prior to randomization), 1 month, and 3 months. The primary endpoint in the trial will be change in self-reported PA minutes from baseline to 3 months. Secondary endpoints will include changes in TPB constructs and quality of life. It is hypothesized that the group receiving the YACS PA guidebook (TARG) will report a greater increase in PA minutes compared to the group receiving Canada's PA guidelines (CPAG).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cancer in Alberta, Canada
* Still living in Alberta, Canada
* Read English

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effects of Targeted Versus Generic Print Materials | One Year
  Behaviour Change

CONTACTS AND LOCATIONS:
Locations (1):
- Behaviour Medicine Laboratory, Edmonton, Alberta, Canada